CLINICAL TRIAL: NCT00669981
Title: Cognitive-Behavioral Couples Therapy for Posttraumatic Stress Disorder
Brief Title: Effectiveness of Cognitive Behavioral Couples Therapy for Post-traumatic Stress Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Candice Monson, Professor & Director of Clinical Training, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH076813 (NIH); R34MH076813 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Post-traumatic Stress Disorder
Keywords: PTSD; Relationship Distress; Couple Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive immediate cognitive behavioral couples therapy for PTSD.
  Interventions: Behavioral: Cognitive behavioral couples therapy for post-traumatic stress disorder (CBCT for PTSD)
- 2 (Active Comparator): Participants will receive delayed cognitive behavioral couples therapy for PTSD after a 3-month waitlist period.
  Interventions: Behavioral: Cognitive behavioral couples therapy for post-traumatic stress disorder (CBCT for PTSD)

INTERVENTIONS:
Behavioral: Cognitive behavioral couples therapy for post-traumatic stress disorder (CBCT for PTSD) — CBCT for PTSD is a 15-session manualized couples therapy that aims to both decrease individual PTSD symptoms and improve dyadic functioning.

SUMMARY:
This study will evaluate the effectiveness of cognitive behavioral couples therapy designed for post-traumatic stress disorder in reducing symptoms of post-traumatic stress disorder and in improving relationship functioning.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is a highly prevalent and disabling disorder that affects about 7.7 million adults in the United States. PTSD can develop after someone experiences a particularly distressing event that may involve the threat of or actual physical harm. Common symptoms of PTSD include avoidance of situations or cues that may act as reminders of the event, reoccurring flashbacks of the event, loss of interest in previously enjoyed activities, and numbing of emotions. Additionally, PTSD is often associated with far-reaching and devastating interpersonal relationship problems that can maintain or aggravate other PTSD symptoms. These interpersonal problems can also interfere with successful treatment delivery, so addressing such problems is important for improving treatment compliance, effectiveness, and long-term success. Cognitive behavioral therapy (CBT) is a type of psychotherapy that teaches ways to modify thoughts and behaviors that contribute to PTSD. CBT that is adapted for couples in which one partner has PTSD may be the most effective means of decreasing individual PTSD symptoms and improving the couple's relationship. This study will evaluate the effectiveness of cognitive behavioral couples therapy (CBCT) for PTSD in reducing symptoms of PSTD and in improving relationship functioning for couples in which one partner has PTSD.

Participation in this study will last 8 months. All participants will undergo baseline assessments that will include an interview about exposure to traumatic events, PTSD symptoms, mental health problems, and substance use; self-report questionnaires about mood, social and leisure activities, and relationships; and a brief video-recorded communication session as a couple. Eligible participants will then be assigned randomly to receive immediate CBCT for PTSD or delayed CBCT for PTSD. Participants in the delayed treatment group will receive active treatment after a 3-month waitlist period. CBCT for PTSD will include fifteen 75-minute couples therapy sessions, occurring twice weekly for 3 weeks and weekly for the remaining 9 weeks of treatment. Sessions will follow manual-based couples therapy and will aim to both decrease individual PTSD symptoms and enhance dyadic functioning. After each session, participants will also complete out-of-session practice assignments that will include completing worksheets and practicing skills taught in therapy sessions.

Participants receiving immediate CBCT for PTSD will undergo subsequent assessments at mid-treatment, end of treatment, and 3 months after the end of treatment. Participants receiving delayed treatment will undergo assessments 1 and 3 months into the wait-list period and at the end of treatment. Assessments will include questions about PTSD and mental health symptoms, alcohol and substance use, intimate relationship functioning, and family and social activities. Participants will repeat the communication session after the end of treatment for the group receiving immediate therapy and at the end of the wait-list period for the delayed treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of PTSD
* An intimate partner willing to participate in treatment

Exclusion Criteria:

* Both partners have PTSD
* Either partner with substance dependence not in remission for at least 3 months before study entry, current uncontrolled bipolar or psychotic disorder, or severe cognitive impairment
* Couple currently experiencing severe intimate aggression or a desire to separate or end their intimate relationship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale | Measured at pre-treatment, mid-treatment, post-treatment, and 3-month follow-up

SECONDARY OUTCOMES:
Dyadic Adjustment Scale | Measured at pre-treatment, mid-treatment, post-treatment, and 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Candice M. Monson, PhD, Principal Investigator — Toronto Metropolitan University
Locations (2):
- VA Boston Healthcare System, Boston, Massachusetts, United States
- Ryerson University, Toronto, Ontario, Canada

REFERENCES:
- [Background] Monson CM, Schnurr PP, Stevens SP, Guthrie KA. Cognitive-Behavioral Couple's Treatment for posttraumatic stress disorder: initial findings. J Trauma Stress. 2004 Aug;17(4):341-4. doi: 10.1023/B:JOTS.0000038483.69570.5b. PMID 15462542
- [Background] Monson CM, Fredman SJ, Adair KC. Cognitive-behavioral conjoint therapy for posttraumatic stress disorder: application to operation enduring and Iraqi Freedom veterans. J Clin Psychol. 2008 Aug;64(8):958-71. doi: 10.1002/jclp.20511. PMID 18613094
- [Derived] Monson CM, Fredman SJ, Macdonald A, Pukay-Martin ND, Resick PA, Schnurr PP. Effect of cognitive-behavioral couple therapy for PTSD: a randomized controlled trial. JAMA. 2012 Aug 15;308(7):700-9. doi: 10.1001/jama.2012.9307. PMID 22893167